CLINICAL TRIAL: NCT00336349
Title: A Study of Intra-dermal Injection of Botulinum Toxin Type A for the Diabetic Neuropathic Foot Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Allergan (Industry)
Responsible Party: Chaur-Jong Hu, Department of Neurology, Taipei Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TMUH20060504
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus; Neuropathic Pain
Keywords: diabetes mellitus; neuropathic pain
MeSH Terms: conditions — Diabetes Mellitus; Neuralgia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Botulinum Toxin Type A

SUMMARY:
Effective treatment of neuropathic foot pain in diabetic patients is very important to improve their quality of life. There are many medications used to reduce the diabetic neuropathic pain, including anticonvulsants, anti-depressants or analgesics, but none is universally satisfied. A few previous studies employing BOTOX® i.d. injection for control of trigeminal neuralgia, post-herpes neuralgia indicate that BOTOX® was effective in controlling neuropathic pain. Intradermal injection of BOTOX® to the dorsum of the foot in diabetics should be effective in controlling diabetes-associated polyneuropathic pain of the foot.

DETAILED DESCRIPTION:
Design: The present study is a single-center, randomized, double-blinded, cross-over study of BOTOX® in diabetic neuropathic foot pain.

Pain Assessment: Subjective intensity of neuropathic pain was rated by a 100 mm visual analogue scale (VAS, 0 = no pain, 100 = unbearable pain). To assess the somatosensory effect of botulinum toxin, we also performed aserial somatosensory evaluations upon bilateral medial (L5 dermatome) and lateral (S1 dermatome) dorsum of the feet, and bilateral medial calves (L4 dermatome). Tactile threshold (TT) values of were assessed by von Frey filament, applied in an ascending and descending order of magnitude. The force required to bend the filaments was converted to log units for further comparison. Pain threshold (PT) to static mechanical stimuli was also determined by von Frey filament upon the above test sites to evaluate the severity of cutaneous allodynia. All subjects underwent the subjective pain rating and somatosensory evaluations (TT and PT) at baseline and each follow-up stage.

Treatment: Treatments will consist of intradermal (i.d). injections of BOTOX® after topical anesthesia over randomly selected 15 patients and saline placebo over the other 15 patients. Dose will be 0.5-1U/cm2 BOTOX®, at total dose of 50 U/foot. A follow-up visit and assessment will be performed at 1, 4 8, 12 weeks following treatment during which the previous tests will be repeated. A cross-over of injection in the Botox group and saline group will be taken at the 12th week and then repeat the assessments at 1, 4, 8, 12 weeks.

Analysis: Comparison between treated feet and non-treated feet based on QVAS and pain sensitivity test and life quality questionnaire by chi-square analysis.

The summary of proposal is as below. Botox: 1. intradermal injection after Topical anesthesia, EMLA 2. 1 cc syringe with 30-gauge needle 3. 50 U/foot 4. 12 points/foot (3×4) A total of 30 cases (15 Botox group, 15 saline group and cross-over 12 weeks later)

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes with medication for diabetes> 3 years (established diagnosis, HbA1C<10% )
2. symptomatic polyneuropathy (stocking distribution and tingling pain)
3. stable but not satisfactory effects of drugs for diabetic neuropathic foot pain (stable effects of medication for over 6 months)
4. fitness of polyneuropathy on Nerve Conduction Velocity (NCV) criteria
5. willing and able to give written informed consent.
6. willing and able to complete the entire study course and comply with study directions.

Exclusion Criteria:

1. Injection not possible due to physiologic barriers.
2. Subject is pregnant or lactating.
3. Females of childbearing age who are not using a reliable method of avoiding pregnancy.
4. Significant medical or psychiatric disease.
5. Any condition that may put the subject at increased risk with exposure to BOTOX®, including
6. diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function.
7. Use of aminoglycoside antibiotics, curare-like agents, or other agents that might interfere with neuromuscular function.
8. Acute medication overuse in the investigator's best judgment.
9. Alcohol or drug abuse.
10. Heavy smokers
11. Infection or skin problems at any of the injection sites.
12. Known allergy or sensitivity to the study medications or its components.
13. Injections of anesthetics or steroids into the study targeted muscles within one month prior to the day of injection
14. Concurrent participation in another clinical trial within 30 days of the beginning of this study.
15. Previous use of botulinum toxin. (Types A or B)
16. Profound atrophy or excessive weakness of the muscles in the target area(s) or injection.
17. Evidence of peripheral artery occlusion
18. Evidence of liver or renal function impairment
19. Evidence old stroke

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
VAS of pain

SECONDARY OUTCOMES:
SF36 for life quality
sleep quality
blood flow of feet

CONTACTS AND LOCATIONS:
Overall Officials: Chaur-Jong Hu, MD, Principal Investigator — Department of Neurology, Taipei Medical University Hospital, Taipei, Taiwan
Locations (1):
- Chaur-Jong Hu, Taipei, Taiwan